CLINICAL TRIAL: NCT00937391
Title: Open-label, Multi-center, Two-stage, Age Stratified, Pharmacokinetic, Safety, and Efficacy Study in Children 2 Months to < 2 Years of Age Undergoing Magnevist Injection Enhanced MRI
Brief Title: Contrast-enhanced MRI in Children 2 Months to <2 Years
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 91784; 2009-013081-17 (EudraCT Number); 312046 (Other: company internal)
Record Dates: First submitted 2009-07-10; First posted 2009-07-13 (Estimated); Results first posted 2011-10-13 (Estimated); Last update posted 2015-11-18 (Estimated); Status verified 2015-10

CONDITIONS: Magnetic Resonance Imaging
Keywords: MRI agents; Magnevist
MeSH Terms: interventions — Gadolinium DTPA

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Gadopentetate dimeglumine (Magnevist, BAY86-6661) (Experimental): For stage 1: Participants received an IV injection of 0.05 mmol/kg Body Weight (BW) (0.1 mL/kg BW) Magnevist. Upon completion of the MR imaging, the participants received another injection of 0.05 mmol/kg for a total cumulative dose of 0.1 mmol/kg BW (0.2 mL/kg BW). For stage 2: Participants received the optimal efficacious dose established in Stage 1 as a single IV injection of Magnevist Injection (0.1 mmol/kg BW (0.2 mL/kg BW)).
  Interventions: Drug: Gadopentetate dimeglumine (Magnevist, BAY86-6661)

INTERVENTIONS:
Drug: Gadopentetate dimeglumine (Magnevist, BAY86-6661) — For stage 1: Participants received an IV injection of 0.05 mmol/kg Body Weight (BW) (0.1 mL/kg BW) Magnevist. Upon completion of the MR imaging, the participants received another injection of 0.05 mmol/kg for a total cumulative dose of 0.1 mmol/kg BW (0.2 mL/kg BW). For stage 2: Participants received the optimal efficacious dose established in Stage 1 as a single IV injection of Magnevist Injection (0.1 mmol/kg BW (0.2 mL/kg BW)).

SUMMARY:
The purpose of this study is to determine pharmacokinetics, safety and efficacy of Magnevist in children 2 months to < 2 years of age

DETAILED DESCRIPTION:
Safety issues are addressed in the AE section

ELIGIBILITY:
Inclusion Criteria:

* Age: 2 months to < 2 years (23 months)
* Participants (male/female) who are scheduled to undergo gadolinium-enhanced MRI
* Able to comply with the study procedures

Exclusion Criteria:

* Clinical unstable participants (eg, intensive care unit)
* Renal Insufficiency
* Participants undergoing chemotherapy </= 48 hours prior to and up to 24 hours after the administration of Magnevist.

Ages: 2 Months to 23 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 54 (Actual)
Dates: Start 2010-01; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (13):
- United States (9):
  - San Diego, California
  - Aurora, Colorado
  - Chicago, Illinois
  - Iowa City, Iowa
  - Kansas City, Missouri
  - St Louis, Missouri
  - Akron, Ohio
  - Hershey, Pennsylvania
  - Houston, Texas
- Germany (4):
  - Dresden, Saxony
  - Halle, Saxony-Anhalt
  - Kiel, Schleswig-Holstein
  - Jena, Thuringia

REFERENCES:
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe — http://www.clinicaltrialsregister.eu/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The date of the first participant, first visit was 21 Jan 2010. The date of the last participant, last visit was 09 Sep 2010. The date of the Blinded Read for Stage 1 was 27 Apr 2010. the date of the Blinded Read for Stage 2 was 08 Sep 2010
Pre-assignment Details: A subject was enrolled in EITHER Stage 1 or Stage 2 and not both. Overall for both stages, 61 participants were Screened, 7 were Screen Failures, and 54 participants were enrolled and treated of which 53 participants completed the study (20 unique participants in Stage 1 and 33 unique participants in Stage 2)
Groups:
- Gadopentetate Dimeglumine (Magnevist, BAY86-6661): For Stage 1: participants received an IV injection of 0.05 mmol/kg Body Weight (BW) (0.1 mL/kg BW) Magnevist. Upon completion of the MR imaging, the participants received another injection of 0.05 mmol/kg for a total cumulative dose of 0.1 mmol/kg BW (0.2 mL/kg BW). For Stage 2: Another group of participants received the optimal efficacious dose established in Stage 1 as a single IV injection of Magnevist Injection (0.1 mmol/kg BW (0.2 mL/kg BW)).
Period: Stage 1
Arm/Group | Gadopentetate Dimeglumine (Magnevist, BAY86-6661)
Started | 20
Treated | 20 (Valid for Full Analysis Set (FAS); includes all participants administered Magnevist Injection)
Completed | 20
Not Completed | 0
Period: Stage 2
Arm/Group | Gadopentetate Dimeglumine (Magnevist, BAY86-6661)
Started | 34 (Stage 1 and Stage 2 are independent each enrolling a different set of participants)
Treated | 34 (Valid for Full Analysis Set; participants administered correct Magnevist dose based on body weight)
Completed | 33 (The number completed includes participants within the FAS and Per Protocol Set (PPS))
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Groups:
- Gadopentetate Dimeglumine (Magnevist, BAY86-6661) - Stage 1: Participants received an IV injection of 0.05 mmol/kg Body Weight (BW) (0.1 mL/kg BW) Magnevist. Upon completion of the MR imaging, the participants received another injection of 0.05 mmol/kg for a total cumulative dose of 0.1 mmol/kg BW (0.2 mL/kg BW).
- Gadopentetate Dimeglumine (Magnevist, BAY86-6661) - Stage 2: Participants received the optimal efficacious dose established in Stage 1 as a single IV injection of Magnevist Injection (0.1 mmol/kg BW (0.2 mL/kg BW)).
- Total: Total of all reporting groups
Arm/Group | Gadopentetate Dimeglumine (Magnevist, BAY86-6661) - Stage 1 | Gadopentetate Dimeglumine (Magnevist, BAY86-6661) - Stage 2 | Total
Number analyzed (Participants) | 20 | 34 | 54
Age, Customized [Number; unit: Participants]
  2 to 6 months | 6 | 11 | 17
  6 to 12 months | 6 | 11 | 17
  12 months to 2 years | 8 | 12 | 20
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 13 | 26
  Male | 7 | 21 | 28
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 19 | 33 | 52
  Asian | 1 | 0 | 1
  Multiple | 0 | 1 | 1
Body Weight [Mean (Standard Deviation); unit: kg] | 8.4 (2.6) | 8.0 (2.0) | 8.1 (2.2)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Diagnostic Adequacy - Open-label Clinical Investigators (Per Protocol Set)
Description: A clinical judgment by the open-label Clinical Investigators (CIs) as to whether ("yes") or not ("no") the CI could make a diagnosis from the image.
Time Frame: Within 5 minutes after injection
Population: The first 3 participants of Stage 1 received 2 IV injections of 0.05 mmol/kg body weight (BW), images were obtained after each injection and an assessment made by the CIs as to diagnostic adequacy.
Measure: Number; unit: Participants
Groups:
- Gadopentetate Dimeglumine - Stage 1 (Comb. Image 0.05 mmol/kg): Participants (n=3) received an IV injection of 0.05 mmol/kg Body Weight (BW) (0.1 mL/kg BW) Gadopentetate dimeglumine.
- Gadopentetate Dimeglumine - Stage 1 (Comb. Image 0.1 mmol/kg): Participants received an IV injection of 0.05 mmol/kg Body Weight (BW) (0.1 mL/kg BW) Gadopentetate dimeglumine. Participants received another injection of 0.05 mmol/kg for a total cumulative dose of 0.1 mmol/kg BW (0.2 mL/kg BW).
Arm/Group | Gadopentetate Dimeglumine - Stage 1 (Comb. Image 0.05 mmol/kg) | Gadopentetate Dimeglumine - Stage 1 (Comb. Image 0.1 mmol/kg)
Number analyzed (Participants) | 3 | 3
Participants
  No | 1 | 0
  Yes | 2 | 3

2. Primary Outcome: Dose Determined by Blinded Readers to be Superior for Diagnosis
Description: Dose superiority was a calculation based upon the Blinder Readers' assessment of 4 visualization parameters
Time Frame: Within 5 minutes after injection
Population: Primary analysis set (the first 5 PPS participants in each age group)
Measure: Number; unit: Participants
Groups:
- Gadopentetate Dimeglumine - Stage 1: Participants received an IV injection of 0.05 mmol/kg Body Weight (BW) (0.1 mL/kg BW) Magnevist. Upon completion of the MR imaging, the participants received another injection of 0.05 mmol/kg for a total cumulative dose of 0.1 mmol/kg BW (0.2 mL/kg BW).
Arm/Group | Gadopentetate Dimeglumine - Stage 1
Number analyzed (Participants) | 15
Participants
  Reader 1, 0.05 mmol/kg | 0
  Reader 2, 0.05 mmol/kg | 1
  Reader 3, 0.05 mmol/kg | 6
  Reader 1, 0.1 mmol/kg | 15
  Reader 2, 0.1 mmol/kg | 14
  Reader 3, 0.1 mmol/kg | 9

3. Primary Outcome: Paired-dose Comparison of Number of Participants With Dose Superiority Determined for 4 Lesion Visualization Variables - Blinded Readers
Description: For each participant, the Blinded Reader indicated which dose had better contrast enhancement, better border delineation, clearer internal morphology, and provided more diagnostic information. The dose chosen for 3 or 4 of these variables was the selected dose for that Reader and participant. If each dose was superior on 2 variables, the dose which provided more diagnostic information was selected for that participant. The dose selected for the majority of participants was the dose selected by that Reader; if chosen by 2 or 3 Readers, it was the selected dose.
Time Frame: Within 5 minutes after injection
Population: Primary Analysis Set (the first 5 PPS participants in each age group)
Measure: Number; unit: Participants
Groups:
- Gadopentetate Dimeglumine - Stage 1 (Comb. Image 0.05 mmol/kg): Participants received an IV injection of 0.05 mmol/kg Body Weight (BW) (0.1 mL/kg BW) Gadopentetate dimeglumine.
Arm/Group | Gadopentetate Dimeglumine - Stage 1 (Comb. Image 0.05 mmol/kg) | Gadopentetate Dimeglumine - Stage 1 (Comb. Image 0.1 mmol/kg)
Number analyzed (Participants) | 15 | 15
Participants
  BR 1 - Diagnostic information | 0 | 15
  BR 2 - Diagnostic information | 1 | 14
  BR 3 - Diagnostic information | 6 | 9
  BR 1 - Contrast enhancement | 0 | 15
  BR 2 - Contrast enhancement | 1 | 14
  BR 3 - Contrast enhancement | 7 | 8
  BR 1 - Border delineation | 0 | 15
  BR 2 - Border delineation | 1 | 14
  BR 3 - Border delineation | 6 | 9
  BR 1 - Internal morphology | 0 | 15
  BR 2 - Internal morphology | 1 | 14
  BR 3 - Internal morphology | 6 | 9

4. Primary Outcome: PK Analysis - Total Clearance (CL)
Description: Total clearance is the fraction of the volume of distribution (Vd) which is completely purified per unit of time and depends also on the plasma half-life of the drug.
Time Frame: 20 to 45 min and 4 to 8 hours post injection
Population: PK population (N=44) was based on the Per Protocol Set (PPS) defined for Stage 1 as all participants (n=18) who received the appropriate dose of Magnevist Injection based on kg body weight (BW) and in Stage 2 as those participants (n=26) who received +/- 10% of the appropriate dose based on kg BW and had values for both PK samples
Measure: Median (Full Range); unit: Liters/hour
Groups:
- Gadopentetate Dimeglumine - Stage 1 and 2: For Stage 1: Participants received an IV injection of 0.05 mmol/kg Body Weight (BW) (0.1 mL/kg BW) Magnevist. Upon completion of the MR imaging, the participants received another injection of 0.05 mmol/kg for a total cumulative dose of 0.1 mmol/kg BW (0.2 mL/kg BW). For Stage 2: Participants received the optimal efficacious dose established in Stage 1 as a single IV injection of Magnevist Injection (0.1 mmol/kg BW (0.2 mL/kg BW)).
Arm/Group | Gadopentetate Dimeglumine - Stage 1 and 2
Number analyzed (Participants) | 44
Liters/hour | 1.012 [0.272 to 1.588]

5. Primary Outcome: PK Analysis - Total Clearance (CL)/Body Weight (BW)
Description: CL/BW = total clearance normalized by BW
Time Frame: 20 to 45 min and 4 to 8 hours post injection
Population: as for outcome 4
Measure: Median (Full Range); unit: Liters/hour/kg
Arm/Group | Gadopentetate Dimeglumine - Stage 1 and 2
Number analyzed (Participants) | 44
Liters/hour/kg | 0.129 [0.059 to 0.166]

6. Primary Outcome: PK Analysis - Volume of Distribution at Steady State (Vss)
Description: Vss is an estimate of drug distribution independent of the elimination process and is proportional to the amount of drug in the body versus the drug plasma concentration at steady-state.
Time Frame: 20 to 45 min and 4 to 8 hours post injection
Population: as for outcome 4
Measure: Median (Full Range); unit: Liters
Arm/Group | Gadopentetate Dimeglumine - Stage 1 and 2
Number analyzed (Participants) | 44
Liters | 1.784 [0.68 to 3.11]

7. Primary Outcome: PK Analysis - Volume of Distribution at Steady State (Vss) /Body Weight (BW)
Description: Vss/BW = volume of distribution at steady state normalized by body weight
Time Frame: 20 to 45 min and 4 to 8 hours post injection
Population: as for outcome 4
Measure: Median (Full Range); unit: Liters/kg
Arm/Group | Gadopentetate Dimeglumine - Stage 1 and 2
Number analyzed (Participants) | 44
Liters/kg | 0.232 [0.192 to 0.27]

8. Primary Outcome: PK Analysis - Area Under the Drug Concentration-time Curve (AUC)
Description: AUC = Area under the drug concentration-time curve from administration to infinity
Time Frame: Samples taken 20 to 45 min and 4 to 8 hours post injection. AUC calculated from time of injection to infinity.
Population: as for outcome 4
Measure: Median (Full Range); unit: µmol•hour/Liter
Arm/Group | Gadopentetate Dimeglumine - Stage 1 and 2
Number analyzed (Participants) | 44
µmol•hour/Liter | 777.5 [600.8 to 1686.3]

9. Primary Outcome: PK Analysis - t 1/2
Description: t 1/2 = termination elimination half-life calculated from the area under the drug concentration-time curve from administration to infinity
Time Frame: Samples taken at 20 to 45 min and at 4 to 8 hours post injection; t 1/2 calculated from area under the drug concentration-time curve from administration to infinity
Population: as for outcome 4
Measure: Median (Full Range); unit: hour
Arm/Group | Gadopentetate Dimeglumine - Stage 1 and 2
Number analyzed (Participants) | 44
hour | 1.483 [1.142 to 8.427]

10. Secondary Outcome: Number of Participants With Number of Lesions Detected - Stage 1
Description: BR = blinded reader; CI = clinical investigator; unenh. image = unenhanced image; comb. image= combined unenhanced and enhanced image. The Blinded Readers and the open-label Clinical Investigators determined the number of participants with 0, 1, 2, and 3 or more lesions.
Time Frame: Within 5 minutes after injection
Population: Full analysis set
Measure: Number; unit: Participants
Groups:
- Gadopentetate Dimeglumine - Stage 1 (Unenh. Image): Unenhanced image was taken before given any injection to Participants.
Arm/Group | Gadopentetate Dimeglumine - Stage 1 (Unenh. Image) | Gadopentetate Dimeglumine - Stage 1 (Comb. Image 0.05 mmol/kg) | Gadopentetate Dimeglumine - Stage 1 (Comb. Image 0.1 mmol/kg)
Number analyzed (Participants) | 20 | 20 | 20
Participants
  BR 1 - 0 lesions | 5 | 5 | 5
  BR 2 - 0 lesions | 7 | 6 | 7
  BR 3 - 0 lesions | 8 | 5 | 6
  CI - 0 lesions | 11 | 11 | 11
  BR 1 - 1 lesion | 7 | 7 | 7
  BR 2 - 1 lesion | 8 | 8 | 7
  BR 3 - 1 lesion | 8 | 10 | 9
  CI - 1 lesion | 6 | 6 | 6
  BR 1 - 2 lesions | 5 | 5 | 5
  BR 2 - 2 lesions | 1 | 2 | 2
  BR 3 - 2 lesions | 0 | 1 | 1
  CI - 2 lesions | 1 | 1 | 1
  BR 1 - 3 or more lesions | 3 | 3 | 3
  BR 2 - 3 or more lesions | 4 | 4 | 4
  BR 3 - 3 or more lesions | 4 | 4 | 4
  CI - 3 or more lesions | 2 | 2 | 2

11. Secondary Outcome: Number of Participants With Number of Lesions Detected - Stage 2
Description: as for outcome 10
Time Frame: Within 5 minutes after injection
Population: Full analysis set
Measure: Number; unit: Participants
Groups:
- Gadopentetate Dimeglumine - Stage 2 (Unenh. Image): Unenhanced image was taken before given any injection to Participants.
- Gadopentetate Dimeglumine - Stage 2 (Comb. Image): Participants received the optimal efficacious dose established in Stage 1 as a single IV injection of Magnevist Injection (0.1 mmol/kg BW (0.2 mL/kg BW)).
Arm/Group | Gadopentetate Dimeglumine - Stage 2 (Unenh. Image) | Gadopentetate Dimeglumine - Stage 2 (Comb. Image)
Number analyzed (Participants) | 34 | 34
Participants
  BR 1 - 0 lesions | 13 | 13
  BR 2 - 0 lesions | 12 | 11
  BR 3 - 0 lesions | 14 | 10
  CI - 0 lesions | 17 | 15
  BR 1 - 1 lesions | 18 | 17
  BR 2 - 1 lesions | 15 | 16
  BR 3 - 1 lesions | 11 | 13
  CI - 1 lesions | 15 | 15
  BR 1 - 2 lesions | 1 | 2
  BR 2 - 2 lesions | 5 | 4
  BR 3 - 2 lesions | 3 | 4
  CI - 2 lesions | 0 | 1
  BR 1 - 3 or more lesions | 2 | 2
  BR 2 - 3 or more lesions | 2 | 3
  BR 3 - 3 or more lesions | 6 | 7
  CI - 3 or more lesions | 2 | 3

12. Secondary Outcome: Number of Participants With Quality of Lesion Visualization - Stage 1
Description: BR = blinded reader; CI = clinical investigator. The Blinded Readers and the open-label Clinical Investigators determined the quality of lesion visualization with the unenhanced and the combined image sets based on a 3-point scale (1=excellent - lesion clearly seen and diagnosis possible; 2=fair but adequate - most of lesion seen and diagnosis possible; and 3=poor - lesion barely seen and diagnosis not possible)
Time Frame: Within 5 minutes after injection
Population: Full analysis set
Measure: Number; unit: Participants
Arm/Group | Gadopentetate Dimeglumine - Stage 1 (Unenh. Image) | Gadopentetate Dimeglumine - Stage 1 (Comb. Image 0.05 mmol/kg) | Gadopentetate Dimeglumine - Stage 1 (Comb. Image 0.1 mmol/kg)
Number analyzed (Participants) | 20 | 20 | 20
Participants
  BR 1 - Excellent (1) | 4 | 7 | 9
  BR 2 - Excellent (1) | 3 | 6 | 8
  BR 3 - Excellent (1) | 2 | 3 | 3
  CI - Excellent (1) | 12 | 16 | 20
  BR 1 - Fair but adequate (2) | 16 | 12 | 10
  BR 2 - Fair but adequate (2) | 17 | 14 | 12
  BR 3 - Fair but adequate (2) | 16 | 15 | 15
  CI - Fair but adequate (2) | 4 | 4 | 0
  BR 1 - Poor (3) | 0 | 1 | 1
  BR 2 - Poor (3) | 0 | 0 | 0
  BR 3 - Poor (3) | 2 | 2 | 2
  CI - Poor (3) | 4 | 0 | 0

13. Secondary Outcome: Number of Participants With Quality of Lesion Visualization - Stage 2
Description: as for outcome 12
Time Frame: Within 5 minutes after injection
Population: Full analysis set
Measure: Number; unit: Participants
Arm/Group | Gadopentetate Dimeglumine - Stage 2 (Unenh. Image) | Gadopentetate Dimeglumine - Stage 2 (Comb. Image)
Number analyzed (Participants) | 34 | 34
Participants
  BR 1 - Excellent (1) | 3 | 25
  BR 2 - Excellent (1) | 7 | 25
  BR 3 - Excellent (1) | 5 | 18
  CI - Excellent (1) | 12 | 32
  BR 1 - Fair but adequate (2) | 25 | 8
  BR 2 - Fair but adequate (2) | 27 | 9
  BR 3 - Fair but adequate (2) | 28 | 16
  CI - Fair but adequate (2) | 14 | 2
  BR 1 - Poor (3) | 6 | 1
  BR 2 - Poor (3) | 0 | 0
  BR 3 - Poor (3) | 1 | 0
  CI - Poor (3) | 8 | 0

14. Secondary Outcome: Number of Participants With Quality of Border Delineation - Stage 1
Description: BR = blinded reader; CI = clinical investigator. The Blinded Readers and the open-label Clinical Investigators determined the quality of border delineation based on a 3-point scale (1=excellent - border completely delineated; 2=fair but adequate - some of the border is delineated; and 3=poor - entire or almost the entire border is not delineated) by image set
Time Frame: Within 5 minutes after injection
Population: Full analysis set
Measure: Number; unit: Participants
Arm/Group | Gadopentetate Dimeglumine - Stage 1 (Unenh. Image) | Gadopentetate Dimeglumine - Stage 1 (Comb. Image 0.05 mmol/kg) | Gadopentetate Dimeglumine - Stage 1 (Comb. Image 0.1 mmol/kg)
Number analyzed (Participants) | 20 | 20 | 20
Participants
  BR 1 - Excellent (1) | 4 | 6 | 10
  BR 2 - Excellent (1) | 3 | 6 | 8
  BR 3 - Excellent (1) | 3 | 3 | 4
  CI - Excellent (1) | 12 | 16 | 19
  BR 1 - Fair but adequate (2) | 15 | 13 | 9
  BR 2 - Fair but adequate (2) | 16 | 14 | 12
  BR 3 - Fair but adequate (2) | 13 | 14 | 15
  CI - Fair but adequate (2) | 5 | 4 | 1
  BR 1 - Poor (3) | 1 | 1 | 1
  BR 2 - Poor (3) | 1 | 0 | 0
  BR 3 - Poor (3) | 4 | 3 | 3
  CI - Poor (3) | 3 | 0 | 0

15. Secondary Outcome: Number of Participants With Quality of Border Delineation - Stage 2
Description: as for outcome 14
Time Frame: Within 5 minutes after injection
Population: Full analysis set
Measure: Number; unit: Participants
Arm/Group | Gadopentetate Dimeglumine - Stage 2 (Unenh. Image) | Gadopentetate Dimeglumine - Stage 2 (Comb. Image)
Number analyzed (Participants) | 34 | 34
Participants
  BR 1 - Excellent (1) | 4 | 21
  BR 2 - Excellent (1) | 6 | 17
  BR 3 - Excellent (1) | 8 | 24
  CI - Excellent (1) | 12 | 32
  BR 1 - Fair but adequate (2) | 24 | 12
  BR 2 - Fair but adequate (2) | 28 | 17
  BR 3 - Fair but adequate (2) | 25 | 10
  CI - Fair but adequate (2) | 14 | 2
  BR 1 - Poor (3) | 6 | 1
  BR 2 - Poor (3) | 0 | 0
  BR 3 - Poor (3) | 1 | 0
  CI - Poor (3) | 8 | 0

16. Secondary Outcome: Most Frequent Diagnostic Findings With Unenhanced Images - Stage 1
Description: BR = blinded reader; CI = clinical investigator. The Blinded Readers and the open-label Clinical Investigators determined the most frequent diagnostic findings with the unenhanced images
Time Frame: Within 5 minutes after injection
Population: Full analysis set
Measure: Number; unit: Participants
Arm/Group | Gadopentetate Dimeglumine - Stage 1
Number analyzed (Participants) | 20
Participants
  Reader 1 - No lesion | 4
  Reader 2 - No lesion | 7
  Reader 3 - No lesion | 8
  CI - No lesion | 6
  Reader 1 - Brain lesion | 8
  Reader 2 - Brain lesion | 6
  Reader 3 - Brain lesion | 4
  CI - Brain lesion | 7

17. Secondary Outcome: Most Frequent Diagnostic Findings With Unenhanced Images - Stage 2
Description: as for outcome 16
Time Frame: Within 5 minutes after injection
Population: Full analysis set
Measure: Number; unit: Participants
Groups:
- Gadopentetate Dimeglumine - Stage 2: Participants received the optimal efficacious dose established in Stage 1 as a single IV injection of Magnevist Injection (0.1 mmol/kg BW (0.2 mL/kg BW)).
Arm/Group | Gadopentetate Dimeglumine - Stage 2
Number analyzed (Participants) | 34
Participants
  Reader 1 - No lesion | 13
  Reader 2 - No lesion | 12
  Reader 3 - No lesion | 14
  CI - No lesion | 11
  Reader 1 - Brain lesion | 9
  Reader 2 - Brain lesion | 10
  Reader 3 - Brain lesion | 10
  CI - Brain lesion | 10

18. Secondary Outcome: Overall Number of Participants With Change in Diagnosis From Unenhanced to Combined Images - Stage 1
Description: The Blinded Readers and the open-label Clinical Investigators determined the number of participants with a change in diagnosis from unenhanced to combined images. BR = blinded reader; CI = clinical investigator
Time Frame: Within 5 minutes after injection
Population: Full analysis set
Measure: Number; unit: Participants
Arm/Group | Gadopentetate Dimeglumine - Stage 1 (Comb. Image 0.05 mmol/kg) | Gadopentetate Dimeglumine - Stage 1 (Comb. Image 0.1 mmol/kg)
Number analyzed (Participants) | 20 | 20
Participants
  BR 1 | 6 | 6
  BR 2 | 1 | 0
  BR 3 | 6 | 6
  CI | 4 | 4

19. Secondary Outcome: Overall Number of Participants With Change in Diagnosis From Unenhanced to Combined Images - Stage 2
Description: as for outcome 18
Time Frame: Within 5 minutes after injection
Population: Full analysis set
Measure: Number; unit: Participants
Arm/Group | Gadopentetate Dimeglumine - Stage 2
Number analyzed (Participants) | 34
Participants
  BR 1 | 10
  BR 2 | 6
  BR 3 | 10
  CI | 8

20. Secondary Outcome: Number of Participants With Specific Change in the Diagnosis From Unenhanced to Combined Images - Stage 1
Description: Those participants for whom the diagnosis changed for at least 1 Blinded Reader from unenhanced to combined images are presented for Stage 1. For completeness, the corresponding data for these participants are presented for the open-label Clinical Investigators. BR=Blinded Reader; CI=Clinical Investigator.
Time Frame: Within 5 minutes after injection
Population: Full analysis set
Measure: Number; unit: Participants
Arm/Group | Gadopentetate Dimeglumine - Stage 1 (Comb. Image 0.05 mmol/kg) | Gadopentetate Dimeglumine - Stage 1 (Comb. Image 0.1 mmol/kg)
Number analyzed (Participants) | 20 | 20
Participants
  BR 1 - from "metastasis" to "liver lesion" | 1 | 0
  BR 2 - from "no lesion" to "vascular malformation" | 1 | 0
  BR 3 - from "no lesion" to "vascular malformation" | 2 | 0
  BR 3 - from "no lesion" to "brain lesion" | 1 | 2
  BR 1 - from "vasc. malform." to "vasc. malfrom." | 2 | 2
  BR 1 - from "brain lesion" to "brain lesion" | 2 | 2
  BR 3 - from "brain lesion" to "brain lesion" | 2 | 2
  BR 1 - from "other" to "other" | 1 | 1
  BR 3 - from "other" to "vascular malformation" | 1 | 1
  BR 1 - from "metastasis" to "metastasis" | 0 | 1
  BR 3 - from "liver lesion" to "metastasis" | 0 | 1

21. Secondary Outcome: Number of Participants With Specific Change in the Diagnosis From Unenhanced to Combined Images - Stage 2
Description: Those participants for whom the diagnosis changed for at least 1 Blinded Reader from unenhanced to combined images are presented for Stage 2. For completeness, the corresponding data for these participants are presented for the open-label Clinical Investigators. BR=Blinded Reader; CI=Clinical Investigator
Time Frame: Within 5 minutes after injection
Population: Full analysis set
Measure: Number; unit: Participants
Arm/Group | Gadopentetate Dimeglumine - Stage 2
Number analyzed (Participants) | 34
Participants
  BR 1 - from "no lesion" to "brain lesion" | 1
  BR 2 - from "no lesion" to "other" | 1
  BR 3 - from "no lesion" to "other" | 2
  BR 3 - from "no lesion" to "infectious disorder" | 2
  BR 1 - from "vasc. malform." to "vasc. malform." | 1
  BR 1 - from "inf. disorder" to "inf. disorder" | 1
  BR 1 - from "brain lesion" to "no lesion" | 1
  BR 1 - from "brain lesion" to "inf. disorder" | 1
  BR 1 - from "brain lesion" to "brain lesion" | 4
  BR 2 - from "brain lesion" to "brain lesion" | 1
  BR 3 - from "brain lesion" to "brain lesion" | 2
  BR 2 - from "renal lesion" to "renal lesion" | 1
  BR 3 - from "renal lesion" to "renal lesion" | 1
  BR 3 - from "not assessable" to "other" | 1
  BR 1 - from "other" to "vascular malformation" | 1
  BR 2 - from "other" to "vascular malformation" | 2
  BR 2 - from "other" to "other" | 1
  BR 3 - from "other" to "other" | 2

22. Secondary Outcome: Number of Participants With Diagnostic Confidence - Stage 1
Description: The overall diagnostic confidence of the Blinded Readers and the open-label Clinical Investigators was indicated on a 3-point scale: 1=not confident; 2=confident; and 3=very confident. BR=Blinder Reader; CI=Clinical Investigator
Time Frame: Within 5 minutes after injection
Population: Full analysis set
Measure: Number; unit: Participants
Arm/Group | Gadopentetate Dimeglumine - Stage 1 (Unenh. Image) | Gadopentetate Dimeglumine - Stage 1 (Comb. Image 0.05 mmol/kg) | Gadopentetate Dimeglumine - Stage 1 (Comb. Image 0.1 mmol/kg)
Number analyzed (Participants) | 20 | 20 | 20
Participants
  BR 1 - not confident | 1 | 0 | 0
  BR 2 - not confident | 3 | 0 | 0
  BR 3 - not confident | 2 | 0 | 1
  CI - not confident | 8 | 1 | 0
  BR 1 - confident | 17 | 17 | 17
  BR 2 - confident | 14 | 7 | 6
  BR 3 - confident | 13 | 13 | 10
  CI - confident | 3 | 5 | 1
  BR 1 - very confident | 2 | 3 | 3
  BR 2 - very confident | 3 | 13 | 14
  BR 3 - very confident | 5 | 7 | 9
  CI - very confident | 9 | 14 | 19

23. Secondary Outcome: Number of Participants With Diagnostic Confidence - Stage 2
Description: as for outcome 22
Time Frame: Within 5 minutes after injection
Population: Full analysis set
Measure: Number; unit: Participants
Arm/Group | Gadopentetate Dimeglumine - Stage 2 (Unenh. Image) | Gadopentetate Dimeglumine - Stage 2 (Comb. Image)
Number analyzed (Participants) | 34 | 34
Participants
  BR 1 - not confident | 3 | 0
  BR 2 - not confident | 3 | 1
  BR 3 - not confident | 1 | 0
  CI - not confident | 10 | 0
  BR 1 - confident | 28 | 18
  BR 2 - confident | 23 | 4
  BR 3 - confident | 27 | 8
  CI - confident | 18 | 4
  BR 1 - very confident | 3 | 16
  BR 2 - very confident | 8 | 29
  BR 3 - very confident | 6 | 26
  CI - very confident | 6 | 30

24. Secondary Outcome: Management Based on Unenhanced Images - Stage 1
Description: For Stage 1 based on unenhanced images, the recommended management is presented as determined by the open-label Clinical Investigators.
Time Frame: Within 5 minutes before injection
Population: Full analysis set (only participants for whom information on management was given)
Measure: Number; unit: Participants
Arm/Group | Gadopentetate Dimeglumine - Stage 1
Number analyzed (Participants) | 18
Participants
  biopsy | 1
  surgery | 2
  follow-up | 3
  medical treatment | 2
  imaging | 10

25. Secondary Outcome: Management Based on Unenhanced Images - Stage 2
Description: For Stage 2 based on unenhanced images, the recommended management is presented as determined by the open-label Clinical Investigators.
Time Frame: Within 5 minutes before injection
Population: Full analysis set (only participants for whom information on management was given)
Measure: Number; unit: Participants
Arm/Group | Gadopentetate Dimeglumine - Stage 2
Number analyzed (Participants) | 32
Participants
  follow-up | 2
  imaging | 30

26. Secondary Outcome: Overall Number of Participants With Change in Management From Unenhanced to Combined Images - Stage 1
Description: For Stage 1, the number of participants for whom the recommended management of the open-label Clinical Investigators changed from unenhanced to combined images is presented for both doses.
Time Frame: Within 5 minutes after injection
Population: Full analysis set
Measure: Number; unit: Participants
Arm/Group | Gadopentetate Dimeglumine - Stage 1 (Comb. Image 0.05 mmol/kg) | Gadopentetate Dimeglumine - Stage 1 (Comb. Image 0.1 mmol/kg)
Number analyzed (Participants) | 20 | 20
Participants | 5 | 12

27. Secondary Outcome: Overall Number of Participants With Change in Management From Unenhanced to Combined Images - Stage 2
Description: For Stage 2, the number of participants for whom the recommended management of the open-label Clinical Investigators changed from unenhanced to combined images is presented for the optimal efficacious dose determined in Stage 1.
Time Frame: Within 5 minutes after injection
Population: Full analysis set
Measure: Number; unit: Participants
Arm/Group | Gadopentetate Dimeglumine - Stage 2
Number analyzed (Participants) | 34
Participants | 30

28. Secondary Outcome: Number of Participants With Specific Change in Management From Unenhanced to Combined Images - Stage 1
Description: The actual change in management from unenhanced to combined images recommended by the open-label Clinical Investigators is presented for both doses in Stage 1
Time Frame: Within 5 minutes after injection
Population: Full analysis set
Measure: Number; unit: Participants
Arm/Group | Gadopentetate Dimeglumine - Stage 1 (Comb. Image 0.05 mmol/kg) | Gadopentetate Dimeglumine - Stage 1 (Comb. Image 0.1 mmol/kg)
Number analyzed (Participants) | 20 | 20
Participants
  from "follow-up" to "surgery" | 1 | 1
  from "imaging" to "surgery" | 2 | 3
  from "imaging" to "follow-up" | 0 | 1
  from "imaging" to "imaging" | 1 | 0
  from "imaging" to "other" | 0 | 6
  from "other" to "follow-up" | 1 | 1

29. Secondary Outcome: Number of Participants With Specific Change in Management From Unenhanced to Combined Images - Stage 2
Description: The actual change in management from unenhanced to combined images recommended by the open-label Clinical Investigators is presented in Stage 2 for the optimal efficacious dose determined in Stage 1
Time Frame: Within 5 minutes after injection
Population: Full analysis set
Measure: Number; unit: Participants
Arm/Group | Gadopentetate Dimeglumine - Stage 2
Number analyzed (Participants) | 34
Participants
  from "imaging" to "surgery" | 3
  from "imaging" to "follow-up" | 16
  from "imaging" to "medical treatment" | 3
  from "imaging" to "imaging" | 3
  from "imaging" to "other" | 7

ADVERSE EVENTS:
Arm/Group | Gadopentetate Dimeglumine - Stage 1 | Gadopentetate Dimeglumine - Stage 2
Serious Adverse Events (participants affected / at risk) | 4/20 | 8/34
Other Adverse Events (participants affected / at risk) | 6/20 | 2/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Gadopentetate Dimeglumine - Stage 1 (N=20) | Gadopentetate Dimeglumine - Stage 2 (N=34)
Krabbe's disease (Congenital, familial and genetic disorders) | 0 | 1
Alagille syndrome (Congenital, familial and genetic disorders) | 0 | 1
Congenital aortic anomaly (Congenital, familial and genetic disorders) | 0 | 1
Intestinal cyst (Gastrointestinal disorders) | 0 | 1
Bronchitis (Infections and infestations) | 1 | 0
Bronchopneumonia (Infections and infestations) | 1 | 0
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Intracranial venous sinus thrombosis (Nervous system disorders) | 1 | 0
Motor developmental delay (Nervous system disorders) | 0 | 1
Neurogenic bladder (Renal and urinary disorders) | 1 | 0
Laryngeal stenosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Adenoidectomy (Surgical and medical procedures) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Gadopentetate Dimeglumine - Stage 1 (N=20) | Gadopentetate Dimeglumine - Stage 2 (N=34)
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1
Pyrexia (General disorders) | 3 | 1
Rhinitis (Infections and infestations) | 1 | 0
Convulsion (Nervous system disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less